CLINICAL TRIAL: NCT05770986
Title: Gluteus Maximus Training Using Power's Program in Chronic Mechanical Low Back Pain
Brief Title: Effect of Power's Program of Gluteus Maximus on LBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alshaymaa Abdeldaiem Abdeldaiem Mohammed, Physical therapist at Central hospital of Alkhanka, Qalyubiya, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 012/003955
Record Dates: First submitted 2022-12-03; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain
Keywords: Disability; Gluteus maximus; Low back pain; Power's program
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly allocated to an experimental and a control group as follow: Group A (n= 26) will receive the eight phases of the Powers program plus a conventional treatment of flexibility exercises, hot pack, transcutaneous electrical stimulation (TENS), prone resisted hip extension for 12 sessions (3 sessions per week for 4 weeks). Group B (n= 26) will receive the same conventional treatment only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A ( power's group) (Experimental): Patients will receive the eight phases of the power's program plus a conventional treatment of flexibility exercises, hot pack, transcutaneous electrical stimulation (TENS), prone resisted hip extension for 12 sessions (3 sessions per week for 4 weeks).
  Interventions: Other: Group A
- Group B ( control) (Active Comparator): Patients will receive a conventional treatment of flexibility exercises, hot pack, transcutaneous electrical stimulation (TENS), prone resisted hip extension for 12 sessions (3 sessions per week for 4 weeks).
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — the patient must attain the goal repetitions (and holds when required) at one level before progressing to the next level. The principal investigator will provide extensive education to the patient while progressing through the program. Three resistance bands will be used through the exercise progression; yellow band (low resistance), green band (moderate resistance) to blue band (high resistance). The patient will progress to more advanced level if he/she can sustain the position with high resistance band (blue) for one minute with three isometric holds of each exercise on each limb. three sets for 10 repetitions will be performed) Phases 1-3 of the program are focused on GMax activation. Phases 4- 5 are focused on GMax strength, and the final three phases emphasize functional applications of the GMax during ballistic tasks.
  Other Names: Power's Program
  Arms: Group A ( power's group)
Other: Group B — Flexibility exercises of the back muscles: knee to chest stretch, bridging, stretching exercises for hip flexors, piriformis, adductors and hamstring will be performed, with a hold of position for 30 s and with repetitions (3-5 times). Static stretches will be held for 30 seconds to induce changes in flexibility and will be repeated for three sets. Three sessions of stretching per week will be performed b. Prone resisted hip extension 10 repetitions for two sets. c. Hot pack: for 10 minutes. d. TENS: The electrodes will be placed over the area of most severe pain for 15 minutes.
  Other Names: Control
  Arms: Group B ( control)

SUMMARY:
Low back pain (LBP) is highly prevalent that causes significant pain and disability. Core muscles are important for LBP. One of them is gluteus maximus, but effect of power's program for this muscle and its role in LBP is lacking in literature, so this study aims to study the effect of power's program of gluteus maximus on LBP.

DETAILED DESCRIPTION:
Chronic mechanical low back pain (CMLBP) is a common musculoskeletal dysfunction affecting 53% of Egyptian population and 1.4 to 20.0% worldwide.

which is a major social and economic burden. Patients with CMLBP experience time loss of work and recently became a workforce burden. Giving the fact that back pain is widely prevalent across Egyptian population and by addressing the functional deficits in those patients, Proper physical therapy intervention can help reducing such burden and improve over all work performance. The 'Powers Program' is a recent concept and it had been proven to be effective in improving lower extremity function and biomechanics. Up to the knowledge of the primary investigator, GMax strengthening using this program has not been conducted in patients with CMLBP. Studying this approach may benefit physical therapists by providing an evidence-based approach in treating patients with CMLBP through exercise therapy and improve functional performance of these patients therefore they can return to normal activities faster. Moreover, this study may benefit researchers interested in Gluteus maximus (GMax) muscle strength. We believe that this study may open up more rooms for future research to address such an important issue.

ELIGIBILITY:
Inclusion criteria

* Both sex.
* Age 21-45 years.
* Chronic mechanical liw back pain for more than 3 years.
* Body mass index 18.4-29.9 kg/m^2.

Exclusion criteria

* Back pain due to specific pathology.
* postoperative
* Trauma to lower quadrant with past 6 months.
* Radicular pain. Lumbar instability.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Severity of low back Pain | 1 year
  Using the Arabic version of visual analogue scale (VAS), the patient will mark on a 0-10 graphic rating scale in which the (0) value indicating no pain,

SECONDARY OUTCOMES:
Severity of low back disability | 1 year
  Arabic version of Oswestry Disability Index (ODI):
  Participants will choose the best answer reflecting their condition in each domain of ODI.
Gluteus maximus strength | 1year
  GMax muscle strength assessment, the following procedure will be followed: Patient Position: prone with knee to be tested flexed to 90 degrees Clinician Position: mid-table on the side to be tested. Elbows in full extension and both hands fixed to stabilize the HHD. HHD Position: just proximal to the popliteal fossa of the limb to be tested Standard Command: "Go ahead, push-push push-push-push, and relax" Method of Testing: 2 trials of 5 second duration, isometric contraction.
Single limb triple hop test for distnace: | One year
  Description: The distance a patient will travel when 3 maximal forward hops will be performed in succession.
Single-Limb Crossover Hop Test for Distance | One year
  Description: The distance a patient will travel in seconds when 3 maximal crossover forward hops are performed. Measurement method: The patient will stand on one limb, with the toes on the starting line. The patient will perform 3 consecutive maximal hops as far as possible forward and land on the same limb while alternately crossing over a 15-cm strip on the floor. The distance hopped will be measured (in centimeter) from the starting line to the point where the patient's heel landed after the third hop.

CONTACTS AND LOCATIONS:
Overall Officials: Enas Fawzy, Principal Investigator — professor, department of physical Therapy for musculoskeletal disorders
Locations (1):
- Central hospital of Alkhanka, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No